CLINICAL TRIAL: NCT00708097
Title: Clinical Efficacy of Fluoride Toothpastes Using an in Situ Caries Model
Brief Title: In Situ Caries Efficacy of Fluoride Toothpastes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: T3508565
Record Dates: First submitted 2008-07-01; First posted 2008-07-02 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Caries
Keywords: fluoride; in situ; remineralization; enamel; caries
MeSH Terms: interventions — Fluorides

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- NaF toothpaste(1450 ppmF) (Experimental): Study toothpaste containing 1450 ppm F as NaF and 0.4% carbopol as excipient.
  Interventions: Drug: NaF
- NaF toothpaste (1400 ppmF) (Active Comparator): Study toothpaste containing 1400 ppm F as NaF
  Interventions: Drug: NaF
- NaMFP/NaF toothpaste (1450 ppmF) (Active Comparator): Reference toothpaste containing 1000 ppm F as NaMFP and 450 ppm F as NaF
  Interventions: Drug: NaF; Drug: NaMFP
- NaF toothpaste (675 ppmF) (Active Comparator): Study toothpaste containing 675 ppm F as NaF
  Interventions: Drug: NaF
- Placebo toothpaste (0 ppmF) (Placebo Comparator): Fluoride free placebo toothpaste (0 ppm F)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NaF — Fluoride
  Other Names: Fluoride
  Arms: NaF toothpaste (1400 ppmF); NaF toothpaste (675 ppmF); NaF toothpaste(1450 ppmF); NaMFP/NaF toothpaste (1450 ppmF)
Drug: Placebo — Placebo
  Arms: Placebo toothpaste (0 ppmF)
Drug: NaMFP — Fluoride
  Arms: NaMFP/NaF toothpaste (1450 ppmF)

SUMMARY:
This study is to evaluate the effect of fluoride dentifrices on enamel with artificial caries lesions in an in situ model

DETAILED DESCRIPTION:
In situ models represent an acceptable approach for testing the anti-caries potential of fluoride products. This study is to evaluate the effect of fluoride dentifrice containing 1450 parts per million fluoride (ppm F) on enamel with artificial caries lesions in an in situ model. The study toothpaste containing sodium fluoride (NaF) and 0.4% carbopol will be compared to 4 other dentifrices. Comparator toothpastes include NaF toothpaste (1400 ppm F), NaF toothpaste (675 ppm F), sodium monofluorophosphate (NaMFP) and NaF toothpaste (1450 ppm F) and placebo toothpaste (0 ppm F).

ELIGIBILITY:
Inclusion Criteria:

* Consent:Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Age:Aged between 18 and 80 years.
* Compliance:Understands and is willing, able and likely to comply with all study procedures and restrictions.
* General Health:Good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or physical examination.
* Fluoride:Currently living in the Indianapolis, Indiana area and not taking fluoride supplements for medical reasons
* Dentures: a)Currently wearing a removable mandibular partial denture with sufficient room in both posterior buccal flange areas to accommodate two enamel specimens on each side, four specimens in total - required dimensions 12 x 7 millimeter (mm) per side. b) Willing to have their denture modified to accommodate enamel test specimens and willing and capable of wearing their removable mandibular partial dentures 24 hours per day during the experimental periods
* Dental health: Have no current active caries or periodontal disease that may compromise the study or the health of the subjects and all restorations in a good state of repair
* Salivary flow:Have a salivary flow rate in the range of normal values (unstimulated whole saliva flow rate = 0.2 milliliter (mL)/minute; gum base stimulated whole saliva flow rate = 0.8 mL/minute)

Exclusion Criteria:

* Pregnancy: Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
* Breast-feeding:Women who are breast-feeding.
* Allergy/Intolerance: Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Antibiotics: Currently taking antibiotics or have taken antibiotics in the two weeks prior to the screening visit
* Clinical Study/Experimental Medication: a) Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit.b) Participation in another GSKCH investigational dental product study within 7 days of first study treatment c)Previous participation in this study.
* Substance abuse: Recent history (within the last year) of alcohol or other substance abuse.
* Personnel:a) A member of the site study staff living in same household.b)An employee of the sponsor. c) Any employee of any toothpaste manufacturer or their spouse or family member

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Indiana University School of Dentistry, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two days before the start of each treatment period, participants received a professional dental cleaning of their natural teeth, then brushed at home with the fluoride-free toothpaste.
Groups:
- Sodium Fluoride (NaF) Toothpaste(1450 Parts Per Million(Ppm)F): Participants brushed their natural teeth for one timed minute with NaF and 0.4% carbopol toothpaste (1450ppmF as NaF), followed by rinsing with 10 milliliters (mL) water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days. During the treatment period, participants wore their partial dentures 24-hours a day, except when cleaning their dentures.
- NaF Toothpaste (1400ppmF): Participants brushed their natural teeth for one timed minute with NaF toothpaste (1400ppmF as NaF), followed by rinsing with 10mL water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days. During the treatment period, participants wore their partial dentures 24-hours a day, except when cleaning their dentures.
- Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF): Participants brushed their natural teeth for one timed minute with NaMFP and NaF toothpaste (1450ppmF - 1000ppmF as NaMFP and 450ppmF as NaF), followed by rinsing with 10mL water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days. During the treatment period, participants wore their partial dentures 24-hours a day, except when cleaning their dentures.
- NaF Toothpaste (675ppmF): Participants brushed their natural teeth for one timed minute with sodium fluoride and silica toothpaste (675ppmF as NaF), followed by rinsing with 10mL water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days. During the treatment period, participants wore their partial dentures 24-hours a day, except when cleaning their dentures.
- Placebo Toothpaste (0ppmF): Participants brushed their natural teeth for one timed minute with fluoride free toothpaste (0ppmF), followed by rinsing with 10mL water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days. During the treatment period, participants wore their partial dentures 24-hours a day, except when cleaning their dentures.
Period: Period 1
Arm/Group | Sodium Fluoride (NaF) Toothpaste(1450 Parts Per Million(Ppm)F) | NaF Toothpaste (1400ppmF) | Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Started | 11 | 12 | 12 | 11 | 11
Completed | 11 | 11 | 12 | 9 | 10
Not Completed | 0 | 1 | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 2 | 0
Not completed — Other Reason | 0 | 0 | 0 | 0 | 1
Period: Period 2
Arm/Group | Sodium Fluoride (NaF) Toothpaste(1450 Parts Per Million(Ppm)F) | NaF Toothpaste (1400ppmF) | Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Started | 10 (Due to crossover design, a different set of subjects received this treatment compared to Period 1.) | 12 (Due to crossover design, a different set of subjects received this treatment compared to Period 1.) | 10 (Due to crossover design, a different set of subjects received this treatment compared to Period 1.) | 11 (Due to crossover design, a different set of subjects received this treatment compared to Period 1.) | 10 (Due to crossover design, a different set of subjects received this treatment compared to Period 1.)
Completed | 10 | 11 | 9 | 10 | 10
Not Completed | 0 | 1 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 1 | 0
Period: Period 3
Arm/Group | Sodium Fluoride (NaF) Toothpaste(1450 Parts Per Million(Ppm)F) | NaF Toothpaste (1400ppmF) | Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Started | 9 (Due to crossover design, a different set of subjects received this treatment compared to Period 2.) | 11 (Due to crossover design, a different set of subjects received this treatment compared to Period 2.) | 10 (Due to crossover design, a different set of subjects received this treatment compared to Period 2.) | 10 (Due to crossover design, a different set of subjects received this treatment compared to Period 2.) | 10 (Due to crossover design, a different set of subjects received this treatment compared to Period 2.)
Completed | 9 | 11 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sodium Fluoride (NaF) Toothpaste(1450 Parts Per Million(Ppm)F) | NaF Toothpaste (1400ppmF) | Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Started | 12 (Due to crossover design, a different set of subjects received this treatment compared to Period 3.) | 9 (Due to crossover design, a different set of subjects received this treatment compared to Period 3.) | 10 (Due to crossover design, a different set of subjects received this treatment compared to Period 3.) | 11 (Due to crossover design, a different set of subjects received this treatment compared to Period 3.) | 8 (Due to crossover design, a different set of subjects received this treatment compared to Period 3.)
Completed | 12 | 9 | 10 | 11 | 8
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Sodium Fluoride (NaF) Toothpaste(1450 Parts Per Million(Ppm)F) | NaF Toothpaste (1400ppmF) | Sodium Monofluorophosphate (NaMFP)/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Started | 8 (Due to crossover design, a different set of subjects received this treatment compared to Period 4.) | 9 (Due to crossover design, a different set of subjects received this treatment compared to Period 4.) | 11 (Due to crossover design, a different set of subjects received this treatment compared to Period 4.) | 10 (Due to crossover design, a different set of subjects received this treatment compared to Period 4.) | 12 (Due to crossover design, a different set of subjects received this treatment compared to Period 4.)
Completed | 8 | 9 | 11 | 10 | 12
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants who received at least one of the treatment dentifrices during the study and had at least one safety assessment after using the treatment dentifrice.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Percentage Surface Microhardness Recovery (%SMHR) of Sound Enamel Specimens Exposed to NaF Toothpaste (1450ppmF) and NaF Toothpaste (1400ppmF)
Description: SMH test was used to assess mineral status of partially demineralized enamel specimens using Wilson 2100 Hardness tester. SMH was determined by measuring the length of the indentations of enamel specimens. An increase in the indentation length compared to the baseline indicates softening/demineralization while decrease in the indentation represents rehardening/ remineralization of enamel surface. Percent SMHR was calculated from indentation values of enamel specimens at baseline(B); after intra-oral exposure(R) on Day 14; and after in-vitro demineralization(D) on Day 14 using formula [(D-R)/(D-B)]*100.
Time Frame: Baseline to 14 days
Population: Intent to Treat (ITT) population: All randomized participants who had at least one post baseline efficacy assessment. Missing data was not imputed. Due to drop outs there were differences in the number of participants (N) per treatment group.
Measure: Least Squares Mean (Standard Error); unit: Percentage SMHR
Groups:
- NaF Toothpaste (1450ppmF): Participants brushed their natural teeth for one timed minute with NaF and 0.4% carbopol toothpaste (1450ppmF as NaF), followed by rinsing with 10 mL water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days. During the treatment period, participants wore their partial dentures 24-hours a day, except when cleaning their dentures.
Arm/Group | NaF Toothpaste (1450ppmF) | NaF Toothpaste (1400ppmF)
Number analyzed (Participants) | 50 | 52
Percentage SMHR | 28.31 (5.54) | 26.32 (5.51)
Statistical Analysis 1: Comparison: NaF Toothpaste (1450ppmF) vs NaF Toothpaste (1400ppmF); Null hypothesis considered population means of the treatments in comparison, to be equal with respect to percent SMH. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p = 0.5757, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 1.98, 95% CI 2-sided [-5.00 to 8.97] — Difference is first named treatment minus second named treatment such that a negative difference favors the first named treatment

2. Secondary Outcome: Percentage SMHR of Sound Enamel Specimens Exposed to NaF Toothpaste (1450ppmF), NaF Toothpaste (1400ppmF), NaMFP/NaF Toothpaste (1450ppmF), NaF Toothpaste (675ppmF) and Placebo Toothpaste (0ppmF)
Description: as for outcome 1
Time Frame: Baseline to 14 days
Population: ITT population: All randomized participants who had at least one post baseline efficacy assessment. Missing data was not imputed. Due to drop out there were differences in the number of participants analyzed per treatment group.
Measure: Least Squares Mean (Standard Error); unit: Percentage SMHR
Groups:
- NaF/Carbopol Toothpaste(1450ppmF): Participants brushed their natural teeth for one timed minute with NaF and 0.4% carbopol toothpaste (1450ppmF as NaF), followed by rinsing with 10 mL water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days. During the treatment period, participants wore their partial dentures 24-hours a day, except when cleaning their dentures.
- NaF Toothpaste(1400ppmF): Participants brushed their natural teeth for one timed minute with NaF toothpaste (1400ppmF as NaF), followed by rinsing with 10mL water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days. During the treatment period, participants wore their partial dentures 24-hours a day, except when cleaning their dentures.
- NaMFP/NaF Toothpaste (1450ppmF): Participants brushed their natural teeth for one timed minute with NaMFP and NaF toothpaste (1450ppmF - 1000ppmF as NaMFP and 450ppmF as NaF), followed by rinsing with 10mL water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days. During the treatment period, participants wore their partial dentures 24-hours a day, except when cleaning their dentures.
Arm/Group | NaF/Carbopol Toothpaste(1450ppmF) | NaF Toothpaste(1400ppmF) | NaMFP/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Number analyzed (Participants) | 50 | 52 | 53 | 53 | 51
Percentage SMHR | 28.31 (5.54) | 26.32 (5.51) | 26.13 (5.49) | 25.52 (5.48) | 53.38 (5.52)
Statistical Analysis 1: Comparison: NaF/Carbopol Toothpaste(1450ppmF) vs NaMFP/NaF Toothpaste (1450ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5387, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 2.17, 95% CI 2-sided [-4.79 to 9.14] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: NaF/Carbopol Toothpaste(1450ppmF) vs NaF Toothpaste (675ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4306, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 2.79, 95% CI 2-sided [-4.18 to 9.77] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: NaF/Carbopol Toothpaste(1450ppmF) vs Placebo Toothpaste (0ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = -25.07, 95% CI 2-sided [-32.09 to -18.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: NaF Toothpaste(1400ppmF) vs NaMFP/NaF Toothpaste (1450ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9567, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 0.19, 95% CI 2-sided [-6.71 to 7.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: NaF Toothpaste(1400ppmF) vs NaF Toothpaste (675ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8188, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 0.81, 95% CI 2-sided [-6.14 to 7.76] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: NaF Toothpaste(1400ppmF) vs Placebo Toothpaste (0ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = -27.06, 95% CI 2-sided [-34.03 to -20.08] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: NaMFP/NaF Toothpaste (1450ppmF) vs NaF Toothpaste (675ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8599, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 0.62, 95% CI 2-sided [-6.28 to 7.51] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: NaMFP/NaF Toothpaste (1450ppmF) vs Placebo Toothpaste (0ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = -27.25, 95% CI 2-sided [-34.20 to -20.30] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: NaF Toothpaste (675ppmF) vs Placebo Toothpaste (0ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = -27.87, 95% CI 2-sided [-34.84 to -20.89] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage SMHR of Demineralized Enamel Specimens Exposed to NaF Toothpaste (1450ppmF), NaF Toothpaste (1400ppmF), NaF Toothpaste (675ppmF), NaMFP/NaF Toothpaste(1450ppmF) and Placebo Toothpaste (0ppmF)
Description: as for outcome 1
Time Frame: Baseline to 14 days
Population: ITT population. All randomized participants who had at least one post baseline efficacy assessment. Missing data was not imputed. Due to drop out there were differences in the number of participants analyzed per treatment group.
Measure: Least Squares Mean (Standard Error); unit: Percentage SMHR
Groups:
- NaF Toothpaste(1450ppmF): Participants brushed their natural teeth for one timed minute with NaF and 0.4% carbopol toothpaste (1450ppmF as NaF), followed by rinsing with 10 mL water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days. During the treatment period, participants wore their partial dentures 24-hours a day, except when cleaning their dentures.
Arm/Group | NaF Toothpaste(1450ppmF) | NaF Toothpaste(1400ppmF) | NaMFP/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Number analyzed (Participants) | 50 | 52 | 53 | 53 | 51
Percentage SMHR | 34.62 (2.82) | 36.06 (2.79) | 31.12 (2.77) | 27.15 (2.77) | 11.10 (2.80)
Statistical Analysis 1: Comparison: NaF Toothpaste(1450ppmF) vs NaF Toothpaste(1400ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5451, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = -1.45, 95% CI 2-sided [-6.15 to 3.26] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: NaF Toothpaste(1450ppmF) vs NaMFP/NaF Toothpaste (1450ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1433, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 3.50, 95% CI 2-sided [-1.20 to 8.19] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: NaF Toothpaste(1450ppmF) vs NaF Toothpaste (675ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0020, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 7.47, 95% CI 2-sided [2.78 to 12.16] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: NaF Toothpaste(1450ppmF) vs Placebo Toothpaste (0ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 23.52, 95% CI 2-sided [18.79 to 28.25] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: NaF Toothpaste(1400ppmF) vs NaMFP/NaF Toothpaste (1450ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0373, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 4.94, 95% CI 2-sided [0.29 to 9.59] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: NaF Toothpaste(1400ppmF) vs NaF Toothpaste (675ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0002, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 8.92, 95% CI 2-sided [4.24 to 13.59] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: NaF Toothpaste(1400ppmF) vs Placebo Toothpaste (0ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 24.97, 95% CI 2-sided [20.27 to 29.66] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: NaMFP/NaF Toothpaste (1450ppmF) vs NaF Toothpaste (675ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0925, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 3.98, 95% CI 2-sided [-0.66 to 8.61] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: NaMFP/NaF Toothpaste (1450ppmF) vs Placebo Toothpaste (0ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 20.03, 95% CI 2-sided [15.35 to 24.70] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: NaF Toothpaste (675ppmF) vs Placebo Toothpaste (0ppmF); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 16.05, 95% CI 2-sided [11.36 to 20.74] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Enamel Fluoride Uptake (Sound Enamel Specimens)
Description: Enamel fluoride uptake was determined using the microdrill enamel biopsy technique. The amount of fluoride uptake by enamel was calculated based on the amount of fluoride (F) divided by the area of the enamel cores. The difference between treatments was calculated with respect to fluoride uptake by enamel.
Time Frame: Baseline to 14 days
Population: ITT population:. All randomized participants who had at least one post baseline efficacy assessment. Missing data was not imputed. Due to drop out there are differences in the number of participants analyzed per treatment group.
Measure: Least Squares Mean (Standard Error); unit: micrograms (μg)*F/centimeters(cm)^2]
Groups:
- NaMFP/ NaF Toothpaste (1450ppmF): Participants brushed their natural teeth for one timed minute with NaMFP and NaF toothpaste (1450ppmF - 1000ppmF as NaMFP and 450ppmF as NaF), followed by rinsing with 10mL water for 10 seconds. Participants continued the study brushing/rinsing regimen at home twice daily for 14 days. During the treatment period, participants wore their partial dentures 24-hours a day, except when cleaning their dentures.
Arm/Group | NaF Toothpaste (1450ppmF) | NaF Toothpaste (1400ppmF) | NaMFP/ NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Number analyzed (Participants) | 50 | 52 | 53 | 53 | 51
micrograms (μg)*F/centimeters(cm)^2] | 648.06 (47.10) | 650.07 (46.30) | 541.16 (45.91) | 487.14 (45.86) | 425.59 (46.67)
Statistical Analysis 1: Comparison: NaF Toothpaste (1450ppmF) vs NaF Toothpaste (1400ppmF); Null hypothesis considered population means of the treatments in comparison, to be equal with respect to EFU. Statistical tests were 2-sided with a significance level of 0.05; Test type: Superiority or Other; p = 0.9697, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = -2.01, 95% CI 2-sided [-106.34 to 102.32] — Difference is first named treatment minus second named treatment such that a positive difference favors the first named treatment
Statistical Analysis 2: Comparison: NaF Toothpaste (1450ppmF) vs NaMFP/ NaF Toothpaste (1450ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0440, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 106.90, 95% CI 2-sided [2.92 to 210.87] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: NaF Toothpaste (1450ppmF) vs NaF Toothpaste (675ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0026, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 160.92, 95% CI 2-sided [56.96 to 264.88] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: NaF Toothpaste (1450ppmF) vs Placebo Toothpaste (0ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 222.47, 95% CI 2-sided [117.58 to 327.36] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: NaF Toothpaste (1400ppmF) vs NaMFP/ NaF Toothpaste (1450ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0382, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 108.91, 95% CI 2-sided [5.98 to 211.83] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: NaF Toothpaste (1400ppmF) vs NaF Toothpaste (675ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0021, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 162.93, 95% CI 2-sided [59.68 to 266.18] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: NaF Toothpaste (1400ppmF) vs Placebo Toothpaste (0ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 224.48, 95% CI 2-sided [120.51 to 328.46] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: NaMFP/ NaF Toothpaste (1450ppmF) vs NaF Toothpaste (675ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.3003, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 54.03, 95% CI 2-sided [-48.56 to 156.61] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: NaF Toothpaste (675ppmF) vs Placebo Toothpaste (0ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.2432, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 61.55, 95% CI 2-sided [-42.14 to 165.24] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 10: Comparison: NaMFP/ NaF Toothpaste (1450ppmF) vs Placebo Toothpaste (0ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0289, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 115.58, 95% CI 2-sided [12.02 to 219.13] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Enamel Fluoride Uptake (Demineralized Specimens)
Description: as for outcome 4
Time Frame: Baseline to 14 days
Population: ITT population: All randomized participants with at least one post baseline efficacy assessment. Missing data was not imputed. Due to drop out there are differences in the number of participants analyzed per treatment group.
Measure: Least Squares Mean (Standard Error); unit: μg*F/cm^2
Arm/Group | NaF Toothpaste(1450ppmF) | NaF Toothpaste (1400ppmF) | NaMFP/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF)
Number analyzed (Participants) | 50 | 52 | 53 | 53 | 51
μg*F/cm^2 | 2499.47 (133.46) | 2513.37 (131.09) | 1923.76 (129.91) | 1861.80 (129.78) | 686.18 (132.20)
Statistical Analysis 1: Comparison: NaF Toothpaste(1450ppmF) vs NaF Toothpaste (1400ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.9293, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = -13.90, 95% CI 2-sided [-322.47 to 294.66] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: NaF Toothpaste(1450ppmF) vs NaMFP/NaF Toothpaste (1450ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0003, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 575.71, 95% CI 2-sided [268.24 to 883.17] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: NaF Toothpaste(1450ppmF) vs NaF Toothpaste (675ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 637.67, 95% CI 2-sided [330.30 to 945.03] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: NaF Toothpaste(1450ppmF) vs Placebo Toothpaste (0ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 1813.29, 95% CI 2-sided [1503.03 to 2123.54] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: NaF Toothpaste (1400ppmF) vs NaMFP/NaF Toothpaste (1450ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0002, ANOVA; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 589.61, 95% CI 2-sided [285.31 to 893.92] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: NaF Toothpaste (1400ppmF) vs NaF Toothpaste (675ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 651.57, 95% CI 2-sided [346.44 to 956.70] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: NaF Toothpaste (1400ppmF) vs Placebo Toothpaste (0ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 1827.19, 95% CI 2-sided [1519.78 to 2134.60] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: NaMFP/NaF Toothpaste (1450ppmF) vs NaF Toothpaste (675ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.6874, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 61.96, 95% CI 2-sided [-241.25 to 365.17] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: NaMFP/NaF Toothpaste (1450ppmF) vs Placebo Toothpaste (0ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 1237.58, 95% CI 2-sided [931.46 to 1543.70] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 10: Comparison: NaF Toothpaste (675ppmF) vs Placebo Toothpaste (0ppmF); [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment and period with subject as a random effect; Adjusted Mean Difference = 1175.62, 95% CI 2-sided [869.15 to 1482.10] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: All AEs encountered or spontaneously reported following administration of any investigational product (including washout product), or for up to 5 days after the last administration of investigational product were recorded.
Groups:
- Overall: All participants received all treatments during the study
Arm/Group | NaF Toothpaste(1450ppmF) | NaF Toothpaste (1400ppmF) | NaMFP/NaF Toothpaste (1450ppmF) | NaF Toothpaste (675ppmF) | Placebo Toothpaste (0ppmF) | Overall
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/52 | 0/53 | 0/53 | 0/51 | 0/57
Other Adverse Events (participants affected / at risk) | 3/50 | 1/52 | 3/53 | 4/53 | 1/51 | 10/57
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NaF Toothpaste(1450ppmF) (N=50) | NaF Toothpaste (1400ppmF) (N=52) | NaMFP/NaF Toothpaste (1450ppmF) (N=53) | NaF Toothpaste (675ppmF) (N=53) | Placebo Toothpaste (0ppmF) (N=51) | Overall (N=57)
Gingival erythema (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.